CLINICAL TRIAL: NCT01746992
Title: An Open-label,Multicenter Randomised Study of CTOP/ITE/MTX Compared With CHOP as the First-line Therapy for the New Diagnosed Young Patients With T Cell Non-hodgkin Lymphoma
Brief Title: CTOP/ITE/MTX Compared With CHOP as the First-line Therapy for Newly Diagnosed Young Patients With T Cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, vice director of Department of Hematology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTOP
Record Dates: First submitted 2012-12-04; First posted 2012-12-11 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: ALK-negative Anaplastic Large Cell Lymphoma; Peripherial T Cell Lymphoma,Not Otherwise Specified; Angioimmunoblastic T Cell Lymphoma; Enteropathy Associated T Cell Lymphoma; Hepatosplenic T Cell Lymphoma; Subcutaneous Panniculitis Like T Cell Lymphoma
MeSH Terms: conditions — Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Subcutaneous panniculitis-like T-cell lymphoma | interventions — Cyclophosphamide; Vincristine; Doxorubicin; Prednisone; prednylidene; Ifosfamide; pirarubicin; etoposide phosphate; Etoposide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pirarubicin (Experimental): 3 cycles of CTOP(cyclophosphamide,vincristin,pirarubicin and prednisone),3 cycles of ITE(ifosfamide, pirarubicin, etoposide)and 2 cycles of methotrexate
  Interventions: Drug: Cyclophosphamide 750mg/m2; Drug: Vincristine 1.4mg/m2; Drug: prednisone 60mg/m2; Drug: ifosfamide 2000mg/m2; Drug: pirarubicin 50mg/m2; Drug: pirarubicin 25mg/m2; Drug: Etoposide phosphate 100mg/m2; Drug: methotrexate 1500mg/m2
- doxorubicin (Active Comparator): 8 cycles of CHOP regimen(cyclophosphamide,vincristin,doxorubicin and prednisone)
  Interventions: Drug: Cyclophosphamide 750mg/m2; Drug: Vincristine 1.4mg/m2; Drug: Doxorubicin 50mg/m2; Drug: prednisone 60mg/m2

INTERVENTIONS:
Drug: Cyclophosphamide 750mg/m2 — day 1 in both arms
  Other Names: CTX
Drug: Vincristine 1.4mg/m2 — day 1
  Other Names: VCR
Drug: Doxorubicin 50mg/m2 — day 1
  Other Names: ADM
  Arms: doxorubicin
Drug: prednisone 60mg/m2 — day1-day5
  Other Names: PRED
Drug: ifosfamide 2000mg/m2 — day 22-day 24
  Other Names: IFO
  Arms: pirarubicin
Drug: pirarubicin 50mg/m2 — day 1
  Other Names: THP
  Arms: pirarubicin
Drug: pirarubicin 25mg/m2 — day 22
  Other Names: THP
  Arms: pirarubicin
Drug: Etoposide phosphate 100mg/m2 — day 22-day 24
  Other Names: VP-16
  Arms: pirarubicin
Drug: methotrexate 1500mg/m2 — day 43
  Other Names: MTX
  Arms: pirarubicin

SUMMARY:
T cell lymphoma is a heterogenic malignancy with poor outcome. Five-year PFS and OS of the patients recieved classic CHOP regimen(cyclophosphamide,vincristin,doxorubicin and predisone)is less than 30%.High dose intensive chemotherapy doesn't demonstrate better response. At present, there is no standardized treatment protocol for this kind of lymphoma.

Between 1994 and 1998,the Scotland and Newcastle Lymphoma Group prospectively collected data on newly diagnosed patients with enteropathy associated T-cell lymphoma (EATL)in the Northern Region of England and Scotland,which is a rare and aggressive type of peripheral T-cell lymphoma.The novel regimen IVE/MTX (ifosfamide, vincristine, etoposide/methotrexate)-ASCT was piloted for patients eligible for intensive treatment,followed by auto-stem cell transplantation.Five-years PFS and OS were 52% and 60% respectively, significantly improved compared with the historical group treated with anthracycline-based chemotherapy. The encouraged results were extended to the peripherial T cell lymphoma-non specified(PTCL-nos).

Past studies suggested pirarubicin was more active to the T cell lymphoma than doxorubicin in vitro based on its high concentration in tumor cells. Clinical data also presented equivalent even superior efficacy of pirarubicin with lower toxicity than doxorubicin. The aim of our study is to compare the response and survival rate of CTOP/ITE/MTX (cyclophosphamide, vincristin,pirarubicin and predisone/ ifosfamide, pirarubicin, etoposide/methotrexate) with those of CHOP regimen,looking forward to its superiority in efficacy and safety for the de novo young patients with T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* pathologic verified mature T cell lymphoma,including ALK-negative anaplastic large cell lymphoma,peripherial T cell lymphoma-non specific type,angioimmunoblastic T cell lymphoma,enteropathy associated T cell lymphoma and hepatosplenic T cell lymphoma
* SGOT/SGPT no more than 2 times of UNL
* serum creatinine no more than 1.5 times of UNL
* signed informed consent

Exclusion Criteria:

* woman in pregnancy or lactation
* allergic to any intervention drug
* insuitable to the study due to severe complication
* enrolled to other study during the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 6 months
3-year PFS | 3 years

SECONDARY OUTCOMES:
overall response rate | 6 months
3-year os | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, Shanghai Municipality, China